CLINICAL TRIAL: NCT04722926
Title: Lyon Prosthetic Joint Infection Retrospective Cohort Study
Brief Title: Lyon PJI Retrospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 268
Record Dates: First submitted 2021-01-15; First posted 2021-01-25 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Bone and Joint Infection
Keywords: prosthesis joint infection; relapse
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PJI: Patients having had a PJI
  Interventions: Other: PJI

INTERVENTIONS:
Other: PJI — patients having had a PJI managed at the CRIOAc Lyon, with or without relapse

SUMMARY:
Bone and joint infections (BJI), although infrequent (prevalence of 70 per 100,000 in France), have a significant economic and clinical impact. Between 2008 and 2013, the prevalence of BJI increased and infections involving joint prosthesis (PJI) represent a third of BJI in France. They are most often post-operative and more expensive than native IOAs.

This study aims to describe PJI and understand the failure mechanisms of PJI in order to improve their management.

ELIGIBILITY:
Inclusion Criteria:

* patients having had a PJI between 2018 and 2020

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients having had a PJI between 2018 and 2020 managed at the CRIOAc Lyon
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
rate of PJI | between 2018 and 2020
  proportion of PJI among all BJI
Description of PJI | between 2018 and 2020
  acute/chronic
Description of type of prosthesis PJI | between 2018 and 2020
  number of prosthesis
Description of patients having had a PJI | between 2018 and 2020
  type of patients: age
Description of comorbidities of patients having had a PJI | between 2018 and 2020
  type of comorbidities..
rate of bacteria | between 2018 and 2020
  epidemiologic description of PJI
description of antibiotic used | between 2018 and 2020
  type of antibiotic : name
description of antibiotic treatment | between 2018 and 2020
  duration of antibiotic treatment
description of surgical treatment | between 2018 and 2020
  type of surgery: 1-step exchange, 2- step exchange, DAIR

SECONDARY OUTCOMES:
rate of failure | between 2018 and 2020
  proportion of patients having a failure
description of the failure | between 2018 and 2020
  type of failure : persistence or surinfection and management of failure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.crioac-lyon.fr/